CLINICAL TRIAL: NCT03705637
Title: Evaluation of Liposomal Bipivicaine in Split Thickness Skin Graft Donor Sites in Burn Patients
Brief Title: Liposomal Bupivicaine for Skin Graft Donor Sites in Burn Patients
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Patient population too low to reasonably continue study, pandemic had started at time of cessation, further leading to study discontinuation.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jonathan Friedstat, Instructor of surgery, Harvard Medical School, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MGH2018P001992
Record Dates: First submitted 2018-09-29; First posted 2018-10-15 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Burns; Postoperative Pain
MeSH Terms: conditions — Burns; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exparel Arm (Experimental): 20ml Exparel + 10ml injectable 0.9% NS (30ml) for every 100cm2 of donor site.
  Interventions: Drug: Exparel

INTERVENTIONS:
Drug: Exparel — * Donor sites will receive up to 50mg of 0.25marcaine with epinephrine injected uniformly into the wound.
  * The donor site will also receive one bottle (266mg) of Exparel, diluted to be administered uniformly into the entire donor site, spaced out ever 3-4cm. The dilution will be as follows:
    o 20ml Exparel + 10ml injectable 0.9% NS (30ml) for every 100cm2 of donor site.
  * Injection of local anesthesia will be performed after the donor site has been harvested and is hemostatic. The goal is to provide the maximum time possible for the local anesthetic to work while under anesthesia, so it can benefit the patient and not be administered at the end of the case just prior to extubation.

SUMMARY:
Burn injuries are painful to patients and the sources of pain result from many areas including: the injury itself, wound care, and surgery. Inpatients that require surgical skin grafting is often required and the donor site of a skin graft is quite painful for patients. The investigators try to minimize that pain with local anesthetic as well as a combination of pain medications, the donor site pain lasts for days and is what patients often report as being the most painful part of their burn care.

There has been the development of a new form of local anesthesia that can last up to 72 hours when injected into tissue. Based on encouraging results in the literature in areas outside of burns, this study aims to evaluate whether administration of this medication at the time of surgery can help improve pain for burn patients in the postoperative period.

DETAILED DESCRIPTION:
Patients suffer from pain resulting from the injury, wound care, and surgical treatment of their burns. As a result, they often require considerable amounts of narcotics. Given the concern for opiate addiction and the national opiate crisis the investigators have tried to explore other non-opiate means of pain control. One of the newest methods for pain relief is with liposomal bupivacaine, which can provide local analgesia for up to 72 hours at the site of injection. This medication has been used with good effect in multiple contexts.

Skin graft donor sites are the most painful portion of their surgical treatment and the pain typically is most severe during the first few days after surgery. For this reason, the investigators believe the addition of Exparel to the donor site will help with improved multi-modal pain control, making patients more comfortable. It also may decrease opiate requirements which would be beneficial for burn patients.

Few previous studies have been conducted using Exparel at the donor sites of skin grafted burn patients. One case series compares usage of Exparel from two different institutions, however the sample size at each was relatively small (n=20, 5, respectively). Their findings suggest that Exparel may be an effective way of managing postsurgical donor site pain. Based on these limited data there is a need for more robust studies, which is the motivation for doing this larger evaluation of patients.

The investigators believe that the use of Exparel can decrease pain for patients after surgery, in particular at their skin graft donor sites. The investigators want to conduct this study to evaluate whether Exparel can improve pain control for their patients and decrease their need for opiate narcotics.

ELIGIBILITY:
Inclusion Criteria:

* Burn size ≤15% TBSA
* Anticipated one trip to operating room for single stage excision and grafting
* Total donor site surface area <500cm2
* Opioid naïve prior to admission for treatment of burn
* Patient able to consent
* 18 years or older

Exclusion Criteria:

Medical Exclusions:

* Cardiac arrhythmias
* Heart block
* Pregnancy
* Breast-feeding mothers who will be unable to stop breastfeeding for 8 days post-injection
* Allergy to bupvicaine
* Bradycardia
* Severe liver disease
* Incapacity to consent themselves
* Unlikely to survive burn Burn related exclusions
* Current substance abuse
* On opioids prior to admission
* Burn larger than 15% TBSA
* Prior autografting for this particular burn

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Morphine milligram equivalents (MME) administered after receiving Exparel | 3 weeks after hospital discharge
  Hypothesis: Subjects that receive Exparel will require fewer opioids to control their pain post-operatively (compared to historical controls).

SECONDARY OUTCOMES:
Length of hospital stay | Up to 4 weeks
  Hypothesis: Subjects who receive Exparel will be ready or discharge sooner than historical controls due to improved pain control

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers outside of those directly involved in this study.

REFERENCES:
- [Background] Rice DC, Cata JP, Mena GE, Rodriguez-Restrepo A, Correa AM, Mehran RJ. Posterior Intercostal Nerve Block With Liposomal Bupivacaine: An Alternative to Thoracic Epidural Analgesia. Ann Thorac Surg. 2015 Jun;99(6):1953-60. doi: 10.1016/j.athoracsur.2015.02.074. Epub 2015 Apr 23. PMID 25912739
- [Background] Mehran RJ, Martin LW, Baker CM, Mena GE, Rice DC. Pain Management in an Enhanced Recovery Pathway After Thoracic Surgical Procedures. Ann Thorac Surg. 2016 Dec;102(6):e595-e596. doi: 10.1016/j.athoracsur.2016.05.050. PMID 27847094
- [Background] Dissanaike S, McCauley J, Alphonso C. Liposomal bupivacaine for the management of postsurgical donor site pain in patients with burn injuries: a case series from two institutions. Clin Case Rep. 2017 Dec 5;6(1):129-135. doi: 10.1002/ccr3.1292. eCollection 2018 Jan. PMID 29375852
- [Background] Kaplan RS, Porter ME. How to solve the cost crisis in health care. Harv Bus Rev. 2011 Sep;89(9):46-52, 54, 56-61 passim. PMID 21939127